CLINICAL TRIAL: NCT03227289
Title: Pregnancy Risk Factors Promote Conversion From Neonatal Respiratory Distress Syndrome(NRDS) to Acute Respiratory Distress Syndrome(ARDS) : a Observational Cohort Study
Brief Title: Acute Respiratory Distress Syndrome(ARDS) in Neonates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: ARDS
Record Dates: First submitted 2017-07-12; First posted 2017-07-24 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: ARDS; NRDS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stayed in NRDS: The neonates with NRDS are stayed in NRDS
  Interventions: Other: Stayed in NRDS
- Converted to ARDS: The neonates with NRDS are converted to ARDS
  Interventions: Other: Converted to ARDS

INTERVENTIONS:
Other: Stayed in NRDS — The neonates with NRDS are stayed in NRDS.
  Groups: Stayed in NRDS
Other: Converted to ARDS — The neonates with NRDS are converted to ARDS.
  Groups: Converted to ARDS

SUMMARY:
Acute respiratory distress syndrome in neonates has been defined in 2015. Earlier identification and successful intervention into the potential pregnancy associated risk factors for the conversion from NRDS to ARDS is one of the most important components of ARDS prevention.

DETAILED DESCRIPTION:
Pregnancy risk factors (PRF), such as intrahepatic cholestasis during pregnancy(ICP), hypertensive disorder complicating pregnancy(HDCP) and gestational diabetes mellitus(GDM), are related to NRDS, ARDS and subsequent death. Meantime, it has also been proven that the prevention of PRF reduces the risk of NRDS and ARDS. However, few study reported the relations between PRF and the conversion from NRDS to ARDS, and it also remains unknown whether treating PRF can reduce the progression from NRDS to ARDS.

We have found that PRF were related to the increase and deterioration of NRDS in a Chinese cohort. The aims of the present study were: 1). to report the effects of PRF on the conversion from NRDS to ARDS. 2). to clarify whether PRF treatment could prevention from conversion from NRDS to ARDS in a Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. The gestational age was less than 37 weeks;
2. These neonates were diagnosed with NRDS; The diagnosis of NRDS was based on clinical manifestations and chest X-ray findings. The clinical signs and symptoms of NRDS were respiratory distress, tachypnea, nasal flaring, groan, and cyanosis after birth. The typical X-ray picture of RDS showed a grain shadow, air bronchogram or white lung.
3. informed parental consent has been obtained

Exclusion Criteria:

1. parents' decision not to participate;
2. major congenital anomalies;
3. died or left the neonatal intensive care unit(NICU) within 24 hour.

Ages: 5 Minutes to 28 Days | Sex: All
Age Groups: Child
Study Population: The gestational age was less than 37 weeks;
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
the effects of Pregnancy risk factors (PRF) on the conversion from NRDS to ARDS | within 28 days
  the effects of Pregnancy risk factors (PRF) on the conversion from NRDS to ARDS
clarify whether PRF treatment could prevention from conversion from NRDS to ARDS | within 28 days
  clarify whether PRF treatment could prevention from conversion from NRDS to ARDS

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided